CLINICAL TRIAL: NCT04511663
Title: The Effectiveness of a 2-year Assertive Community Treatment on Schizophrenic Patients in an Urban District of Shanghai
Brief Title: The Effectiveness of Assertive Community Treatment on Schizophrenic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WeiboZhang
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Assertive community treatment; Community rehabilitation
MeSH Terms: conditions — Schizophrenia | interventions — Community Mental Health Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A single-blind method was used, in which all the assessments were independently completed by trained psychiatrists who didn't know the grouping.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): The intervention group received assertive community treatment, in which the team consisted of psychiatrists, nurses, clinical psychologists, social workers, rehabilitation teachers.
  Interventions: Combination Product: Assertive community treatment
- control group (Other): The control group received basic public health services which is regular medical follow-up including symptom and medication evaluation, social function evaluation and physical examination after hospital discharge.
  Interventions: Combination Product: Basic public health services.

INTERVENTIONS:
Combination Product: Assertive community treatment — The intervention team consisted of psychiatrists, nurses, clinical psychologists, social workers, rehabilitation teachers. The specific services provided by the team include individual service plan. Each patient got a comprehensive evaluation within one month to establish treatment goals and individual intervention plan, rehabilitation training, family intervention peer support group, individual psychological counseling and crisis intervention.
  Arms: intervention group
Combination Product: Basic public health services. — The control group received regular medical follow-up including symptom and medication evaluation, social function evaluation and physical examination after hospital discharge. The frequency was once a quarter.
  Arms: control group

SUMMARY:
Assertive community treatment (ACT) is a community-based, patient-centered, and rehabilitation-oriented model based on multidisciplinary service teams. It has been proved to be suitable for the management of patients with severe mental disorder in the community. In this study, we aimed to investigate the effectiveness of ACT in an urban district of Shanghai with a larger sample size and a 24-month duration of follow up. We hypothesized that patients assigned into ACT would show better improvement in psychiatric symptoms and social function.

DETAILED DESCRIPTION:
Assertive community treatment (ACT) is a community-based, patient-centered, and rehabilitation-oriented model based on multidisciplinary service teams. It has been proved to be suitable for the management of patients with severe mental disorder in the community. In this study, we aimed to investigate the effectiveness of ACT in an urban district of Shanghai with a larger sample size and a 24-month duration of follow up. We hypothesized that patients assigned into ACT would show better improvement in psychiatric symptoms and social function.The study protocol was approved by the Institutional Review Board in Shanghai Mental Health Center.

Aim of the study: 1.1 To explore the effectiveness of assertive community treatment in patients with schizophrenia. 1.2 The patients were followed up for 24 months to explore the duration of ACT.

Introduction of the study: Patients who previously diagnosed as schizophrenia according to International Classification of Diseases 10th Revision (ICD-10) in the psychiatric hospitals would receive basic public health service in the community. The selected schizophrenic patients were randomly assigned into intervention group and control group by a computer randomization algorithm. During the following 2 years, the control group received basic public health services in the community while the intervention group received ACT. Clinical assessments were conducted at baseline and every 6 months till the end of the 2-year study. A single-blind method was used, in which all the assessments were independently completed by trained psychiatrists who didn't know the grouping.The Positive and Negative Symptoms Scale (PANSS) and the Personal and Social Performance Scale (PSP) were measured at baseline and every 6 months during the study.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 50 years old;
2. course of disease between 2 and 20 years;
3. living with family members who can function as their caregivers;
4. disease condition was stable and the total score of the Positive and Negative Symptoms Scale (PANSS) is less than 60.

Exclusion Criteria:

1. women during pregnancy;
2. having mental retardation or psychoactive substance-induced mental disorders;
3. having serious physical condition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
PANSS | 6 months
  PANSS（Positive and Negative Syndrome Scale） is a relatively mature assessment tool commonly used in clinical research to assess the severity of schizophrenia symptoms. It consists of a positive symptom subscale (7 items), a negative symptom subscale (7 items) and a general psychopathological symptom subscale (16 items), a total of 30 items.Each item has specific definitions and operational grading criteria. It is divided into 7 grades according to the level of psychopathology (1~7 points). The higher the score, the heavier the symptoms. The total score of PANSS is 30- 210 points, the positive symptom subscale and the negative symptom subscale are 7-49 points, and the general psychopathological symptoms subscale is 16 to 112 points.

SECONDARY OUTCOMES:
PSP | 6 months
  PSP (The Personal and Social Performance Scale) uses a 100-point rating scale to assesses social functioning. A score of 71-100 indicates mild difficulties in social functioning; 31-70 indicates varying degrees of impairment and disability; and 0-30 indicates poor functioning that requires intensive support or supervision. Chinese version of the PSP demonstrated good psychometric characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No